CLINICAL TRIAL: NCT05901896
Title: Temporal Changes in Gut Microbiota of Healthy Adults Before and After Migrating to High Altitude: a Longitudinal Study
Brief Title: Temporal Changes in the Gut Microbiota Before and After Migrating to High Altitude
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Gut Microbiota001
Record Dates: First submitted 2023-05-17; First posted 2023-06-13 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-02

CONDITIONS: Gut Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: The study group consists of five volunteers who originally lived in a plain area. They will be living in a high-altitude region for one year.
  Interventions: Other: there are no intervention
- control group: Five healthy residents living on the high-altitude region , matched 1:1 by age, gender, and race, will serve as control group.
  Interventions: Other: there are no intervention

INTERVENTIONS:
Other: there are no intervention — no intervention

SUMMARY:
This prospective observational cohort study aims to learn about temporal changes in the gut microbiota before and after migrating to high altitudes in healthy participants. The main questions it aims to answer are:

* changes in the gut microbiome before and after migrating to high altitude.
* Do the migrants tend to share similar gut microbiota characteristics with the residents? Participants will detect 16S ribosomal RNA profiles from stool samples. Researchers will compare the residents with the migrants to see if gut microbiota characteristics are similar.

DETAILED DESCRIPTION:
Changes in geographical environment can lead to alterations in the composition of the host's gut microbiota. However, the dynamic process and specific bacterial composition and patterns of change in the microbiota are not yet clear. In this study, the investigators conducted microbial analysis of the gut microbiota based on 16S rRNA amplicon sequencing in five healthy volunteers living in a plain area (Liaocheng City, Shandong Province) before and after their relocation to a high-altitude region (Gangcha County, Qinghai Province). Samples were collected at multiple time points, including 1 month, 3 months, 6 months, and 12 months after relocation, as well as 1 month, 3 months, 6 months, and 12 months after returning to Liaocheng City from Gangcha County. Additionally, a control group consisting of five local healthy individuals from Gangcha County (matched for age, gender, and ethnicity in a 1:1 ratio) was included. Dietary and lifestyle habits were investigated to determine the impact of environmental changes on the gut microbiota. The study aimed to analyze the diversity and abundance changes of the gut microbiota at different time points and identify specific bacterial compositions through clustering analysis.

ELIGIBILITY:
Inclusion criteria:

Volunteers in good health, without any diagnosed chronic diseases or gastrointestinal disorders.

Exclusion criteria:

recent antibiotic use; severe gastrointestinal infections; long-term use of immunosuppressive drugs or other medications that may impact the gut microbiota; history of gastrointestinal surgical interventions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group consists of five volunteers who originally lived in a plain area. They will be living in a high-altitude region for one year. Five healthy residents living on the high-altitude region , matched 1:1 by age, gender, and race, will serve as control group.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
the bacterial composition difference using 16S rRNA sequencing 1 | one month after relocation
  Alpha and beta diversity were calculated based on the rooted phylogenetic tree. Read classification to taxonomic profiles at four levels e.g., phylum, family, genus and species was compared between baseline and one month after relocation.
the bacterial composition difference using 16S rRNA sequencing 2 | three month after relocation
  Alpha and beta diversity were calculated based on the rooted phylogenetic tree. Read classification to taxonomic profiles at four levels e.g., phylum, family, genus and species was compared between baseline and three month after relocation.
the bacterial composition difference using 16S rRNA sequencing 3 | six month after relocation
  Alpha and beta diversity were calculated based on the rooted phylogenetic tree. Read classification to taxonomic profiles at four levels e.g., phylum, family, genus and species was compared between baseline and six month after relocation.
the bacterial composition difference using 16S rRNA sequencing 4 | twelve month after relocation
  Alpha and beta diversity were calculated based on the rooted phylogenetic tree. Read classification to taxonomic profiles at four levels e.g., phylum, family, genus and species was compared between baseline and twelve month after relocation.

SECONDARY OUTCOMES:
the bacterial composition difference using 16S rRNA sequencing 5 | one month after returning to Liaocheng City from Gangcha County.
  Alpha and beta diversity were calculated based on the rooted phylogenetic tree. Read classification to taxonomic profiles at four levels e.g., phylum, family, genus and species was compared between baseline and one months after returning to Liaocheng City from Gangcha County.
the bacterial composition difference using 16S rRNA sequencing 6 | three month after returning to Liaocheng City from Gangcha County.
  Alpha and beta diversity were calculated based on the rooted phylogenetic tree. Read classification to taxonomic profiles at four levels e.g., phylum, family, genus and species was compared between baseline and three months after returning to Liaocheng City from Gangcha County.
the bacterial composition difference using 16S rRNA sequencing 7 | six month after returning to Liaocheng City from Gangcha County.
  Alpha and beta diversity were calculated based on the rooted phylogenetic tree. Read classification to taxonomic profiles at four levels e.g., phylum, family, genus and species was compared between baseline and six months after returning to Liaocheng City from Gangcha County.
the bacterial composition difference using 16S rRNA sequencing 8 | twelve month after returning to Liaocheng City from Gangcha County.
  Alpha and beta diversity were calculated based on the rooted phylogenetic tree. Read classification to taxonomic profiles at four levels e.g., phylum, family, genus and species was compared between baseline and twelve months after returning to Liaocheng City from Gangcha County.

CONTACTS AND LOCATIONS:
Locations (1):
- Liaocheng people's hospital, Liaocheng, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided